CLINICAL TRIAL: NCT00578838
Title: Magnetic Resonance Study of Liver in Chemotherapy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-082
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 25 patients with metastatic colorectal cancer. Each patient will have 4 MR exams: prior to or within one week of the start of the chemotherapy regimen, one after 6 weeks of chemotherapy, a third after completion of chemotherapy (between 12 and 24 weeks post-initiation of chemotherapy) and a long term followup study at least 4 months after the completion of chemotherapy.
  Interventions: Other: Magnetic Resonance
- 2: 25 patients with non-metastatic colorectal cancer. Each patient will have 4 MR exams: prior to or within one week of the start of the chemotherapy regimen, one after 6 weeks of chemotherapy, a third after completion of chemotherapy (between 12 and 24 weeks post-initiation of chemotherapy) and a long term followup study at least 4 months after the completion of chemotherapy.
  Interventions: Other: Magnetic Resonance
- 3: 11 healthy volunteers, who will also undergo two scans 2-3 weeks apart.
  Interventions: Other: Magnetic Resonance

INTERVENTIONS:
Other: Magnetic Resonance — Patients each will undergo 4 MR examinations as part of this research study.
  Groups: 1; 2
Other: Magnetic Resonance — You will have two MR exams on two different days. There will be no injection of contrast material. An MR exam requires about 1 hour. The second MR exam will take place 2-3 weeks after the first one. This second MR exam will take about 1 hour and will look at whether the results from the MR exams are reliable and repeatable.
  Groups: 3

SUMMARY:
The purpose of this study is to see whether magnetic resonance (MR) techniques can detect changes caused by chemotherapy in the livers of patients who have been treated for colorectal cancer. Some patients who undergo chemotherapy for colorectal cancer may experience side-effects in their livers. These side effects may influence further treatment options. If this study finds that MR techniques detect changes in the liver due to chemotherapy, then MR methods may eventually be used to help patients and physicians plan further treatment.

DETAILED DESCRIPTION:
Each patient will have 4 MR exams: prior to or within one week of the start of the chemotherapy regimen, one after 6 weeks of chemotherapy, a third after completion of chemotherapy (between 12 and 24 weeks post-initiation of chemotherapy) and a long term followup study at least 4 months after the completion of chemotherapy. Normal volunteers will be recruited and studied by MR for comparison to patient data.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* 21 years of age or older.
* Histologically confirmed diagnosis of colorectal carcinoma (patients only).
* Resected primary colorectal cancer and no metastatic disease or primary colorectal cancer with no metastatic disease and planned resection after neo-adjuvant chemotherapy or metastatic colorectal carcinoma considered by the attending physician to have resectable or potentially resectable hepatic metastases (patients only). Each patient will be staged by his/her attending physician in the Department of Medicine or Surgery. Hepatic metastases are considered resectable if they are expected to be completely removable with negative margins by a procedure that leaves behind sufficient liver parenchyma with arterial/portal blood supply, venous drainage and biliary drainage for subsequent regeneration and survival. Potentially resectable indicates that a reduction in tumor size due to chemotherapy could render the tumors resectable.

Exclusion Criteria:

* Inability to cooperate for an MR exam.
* Contraindication to MR:

  * Pacemaker
  * Aneurysmal clips
  * Any ferrous metallic implants which could be deflected by the magnet
  * Metal implants in field of view which could distort the images and spectroscopy data
  * Pregnant women
  * Age and mental status wherein he/she is unable to cooperate for MR study
* Patients who are considered to have unresectable hepatic metastases will be excluded. Hepatic metastases are considered unresectable if their removal would leave behind insufficient liver parenchyma for subsequent regeneration and survival. In addition, hepatic metastases are considered unresectable if their removal would be expected to leave behind residual disease (positive margins). Also, patients are considered unresectable if they have any comorbid conditions which would jeopardize successful recovery from hepatic resection.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be a total of 20 patients with metastatic colorectal cancer, 20 patients with non-metastatic colorectal cancer and 11 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2006-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To determine whether magnetic resonance techniques can detect changes in normal liver morphology and metabolism caused by chemotherapy in patients with colorectal cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Zakian, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org